CLINICAL TRIAL: NCT03910296
Title: Acceptance and Commitment Therapy (ACT) - Based Treatment Development for Cancer Patients Treated for Pain
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, MiryamYusufov, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 19-035
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acceptance & Commitment Therapy: * Acceptance & Commitment Therapy (ACT) use acceptance, mindfulness, commitment, and behavior change strategies to increase psychological flexibility.
  * Each subject will participate for 6 sessions of Acceptance & Commitment Therapy (ACT).
  * ACT trains patients to reframe their unpleasant, negative, private events while encouraging personal values.
  Interventions: Behavioral: Acceptance & Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance & Commitment Therapy — ACT is a unique, third-wave therapy that uses metaphors and experiential exercises to encourage contact with previously avoided thoughts, feelings, and behaviors.

SUMMARY:
The purpose of this research study is to develop a psychological treatment for patients with cancer, focused on the psychological symptoms they experience during opioid therapy.

DETAILED DESCRIPTION:
This research study is a treatment development study, which is the first time investigators are developing this psychological intervention in patients with cancer, on opioid therapy. This study is being conducted to develop a psychological intervention designed specifically for individuals with cancer. The purpose of this study is to determine how practical this intervention is, to determine patient satisfaction, and test the study procedures.

ELIGIBILITY:
Inclusion Criteria:

* must be at least 18 years of age
* speak and comprehend English sufficiently to be able to complete the study procedures and participate in psychotherapy in English
* have been diagnosed with cancer
* have an estimated survival time ≥6 months (as approximated by palliative care clinic staff)
* score ≥4 on the Opioid Risk Tool (Webster & Webster, 2005) with psychosocial distress as one of the positive items.

Exclusion Criteria:

* untreated bipolar disorder
* untreated psychotic disorders
* untreated borderline personality disorder
* have an estimated survival time ≤6 months (as approximated by clinic staff).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All potentially eligible patients will be identified through the DFCI ambulatory palliative care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Study feasibility | 2 years
  Defined by participants' completion of 80% of measures

SECONDARY OUTCOMES:
Intervention acceptability | 2 years
  Defined by participant responses on the semi-structured qualitative interviews, upon treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Miryam Yusufov, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation